CLINICAL TRIAL: NCT00901537
Title: Phase I Study of Azacitidine in Combination With Cisplatin in Patients With Recurrent or Metastatic Non-small Cell Lung Cancer or Squamous Cell Carcinoma of the Head and Neck
Brief Title: Azacitidine and Cisplatin in Patients With Advanced Lung or Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor terminated due to no enrollments within last 4 months.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Chung-Tsen Hsueh, MD PhD, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 58358; IND 105076 (IND Exempt)
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Non-small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck
Keywords: Non-small Cell Lung Cancer; Head and Neck Cancer; Azacitidine; Vidaza; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Azacitidine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacitidine and Cisplatin (Experimental): Every 4 weeks, azacitidine is given daily as subcutaneous injection for 5 days from day 1 to day 5, and cisplatin is given as intravenous injection on day 8. The dose of azacitidine will be dose escalated among each group of 3-6 patients, and the dose of cisplatin is fixed.
  Interventions: Drug: Azacitidine and Cisplatin

INTERVENTIONS:
Drug: Azacitidine and Cisplatin — We plan to give azacitidine daily as subcutaneous injection at escalated doses (37, 60, 75, 85, 100 and 110 mg/m2) for 5 days from day 1 to day 5, and give cisplatin 75 mg/m2 as intravenous injection on day 8, every 4 weeks as a cycle.
  Other Names: Vidaza; 5-Azacytidine

SUMMARY:
The standard of care for head and neck and lung cancer includes chemotherapy, radiation and surgery. For patients with cancer of head and neck or lung that recurs after surgery and/or radiation, or has spread to other parts of body, chemotherapy using cisplatin can slow down tumor growth and extend lifespan.

The study drug, azacitidine, can block the ability of some cancer cells to replicate, and has been approved by the Food and Drug Administration for use in myelodysplastic syndrome, which is a slowly developing blood cell-related cancer. In laboratory and animal experiments using head and neck and lung cancer cells, azacitidine has been shown to be a cisplatin "helper", (that is, it makes cisplatin more effective in stopping the growth of head and neck and lung cancer. )

Since the combination of azacitidine and cisplatin has not been used in patients with head and neck or lung cancer, the investigators are performing this study combining azacitidine and cisplatin to find out what effects, good and/or bad, the study drug may have on patients with advanced head and neck or lung cancer. The investigators are doing this study because they would like to find a better treatment for these types of cancer.

DETAILED DESCRIPTION:
Azacitidine will be given with standard dose of cisplatin. At the beginning of the study, three patients will be treated with low dose of azacitidine. If that dose does not cause bad side effects, then the dose will slowly be made higher for new patients who take part in the study.

Patients will receive azacitidine as a once-a-day subcutaneous (under the skin) injection every day from day 1 to day 5 of 28 days in this study. Cisplatin is given intravenously on day 8. This 28-day or 4-week period of time is called a cycle. Cycles are repeated every four weeks for as long as the physician recommends.

During this study, patients will need the following tests and procedures.

* Physical exam - This will be done weekly during first 2 weeks of every 4-week treatment cycle.
* Blood tests for blood counts - These will be done every week.
* Blood tests for kidney function, liver function, and to measure electrolytes - These will be done every week
* Blood samples for research study - This will be done weekly during first cycle, then weekly during the first 2 weeks on the subsequent treatment cycles
* X-rays or scans - These will be done once every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven squamous cell carcinoma of head and neck or non-small cell lung cancer that is either metastatic or has persisted or recurred following definitive surgery and/or radiation therapy, and is not amenable to salvage surgical resection.
* Patients may have received previous chemotherapy and/or biological treatment such as cetuximab, bevacizumab or erlotinib) for the recurrent or metastatic disease. Prior treatment must have been completed at least 28 days (42 days for nitrosoureas or mitomycin C) prior to entering the study and all toxicities must have been resolved. Patients who have received prior treatment with EGFR inhibitor alone such as cetuximab or erlotinib are allowed to enter the study at least 14 days after receiving the last dose of the prior treatment.
* Prior radiation must have been completed at least 28 days before entry into the study and all toxicities must have been resolved (no more than 3000 cGy to fields including substantial marrow).
* Surgery must have been completed at least 28 days 28 days before entry into the study and all complications/adverse events must have been resolved.
* Age >18 years.
* ECOG performance status <2 (Karnofsky >60%).
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function
* Patients must not be planning to receive any other concurrent therapy (i.e. radiation, chemotherapy, immunotherapy, biological therapy or gene therapy) while they are on this study.
* Patients must be able to understand and sign a written informed consent document approved for this trial.
* Women of childbearing potential must have a negative serum pregnancy test prior to azacitidine treatment.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this clinical trial. Patients with asymptomatic brain metastases are allowed. The patient must be stable for 2 weeks after radiotherapy; if the patient is on corticosteroids, the dose of cortico steroids must have been stable for 2 weeks prior to first dose of study treatment, or be in the process of being tapered.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to azacitidine, cisplatin and mannitol or other agents used in study.
* Pregnant or nursing women may not participate in this trial because of the increased risk of fetal harm including fetal death from the chemotherapeutic agents. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients known to be HIV-positive are not eligible because of the potential to confound this study's endpoints.
* No prior malignancy is allowed except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer or other cancer for which the patient has been disease-free for five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and toxicity of azacitidine and cisplatin combination. | weekly for first 4 weeks, then weekly times 2 for every 4 weeks

SECONDARY OUTCOMES:
Determine the biologically effective dose of azacitidine, maximum tolerated dose of azacitidine and cisplatin combination, and tumor response | every 8 weeks for response evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Tsen Hsueh, MD, PhD, Principal Investigator — Loma Linda University Cancer Center
Locations (1):
- Loma Linda University Cancer Center, Loma Linda, California, United States